CLINICAL TRIAL: NCT04821115
Title: Safety and Efficacy of Low-intensity Shockwave Therapy for Peyronie's Disease
Acronym: ONDELA
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Hopital Foch (Other)
Collaborators: Dornier MedTech Systems (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: 2019_0075
Record Dates: First submitted 2021-03-25; First posted 2021-03-29 (Actual); Last update posted 2024-07-31 (Actual); Status verified 2024-07

CONDITIONS: Peyronie Disease; Penile Diseases
MeSH Terms: conditions — Penile Induration; Penile Diseases

STUDY DESIGN:
Who Masked: Participant, Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- Low intensity choc waves therapy (Experimental group) (Experimental): The patients will use the device with a real applicator.
  Interventions: Device: Low intensity choc waves therapy (active applicator)
- Sham group (Sham Comparator): The patients will use the device with a sham applicator. Instead of a focusing lens, the applicator will have an internal foam piece that will dissipate the energy of the shockwave. Hence, the sham applicator will look, feel and sound the same as the active, but no measurable energy is emitted
  Interventions: Device: Sham (sham applicator)

INTERVENTIONS:
Device: Low intensity choc waves therapy (active applicator) — At each of the 4 sessions, 4000 shockwaves will be delivered at level 8 (EFD = 0.133 mJ/mm2), over a period of 15 to 20 minutes. The probe will be applied directly to the plaque, on the flaccid penis. The device will stop automatically after the 4000 shock waves.
  Arms: Low intensity choc waves therapy (Experimental group)
Device: Sham (sham applicator) — At each of the 4 sessions, a sham applicator will be used. The sham applicator has an internal foam pad that disperses the shockwave energy, but is not visible from the outside. The sham applicator will look, feel and sound the same as the active, but no measurable energy is emitted.
  Arms: Sham group

SUMMARY:
Investigation of the effect of Low-intensity extracorporeal shockwave therapy (ESWT) for Peyronie's disease (PD) via a single blind, sham-controlled, randomized clinical trial. Investigators will not be blinded to group assignments, but penile curvature will be assessed from coded patient pictures by a blinded assessor.

ELIGIBILITY:
Inclusion Criteria:

* ≥18 years old male,
* Untreated Peyronie's disease (excepted oral therapy) (wash out: at least 1 month),
* Single axis penile curvature in erection at 20 - 90 degrees at baseline,
* Dorsal or lateral penile plaque,
* Able and willing to perform ESWT self-treatment under supervision,
* Able to understand and complete patient questionnaires,
* Having sign an informed consent form prior to any study specific procedure,
* Being covered by a national health insurance

Exclusion Criteria:

* Congenital penile deformity,
* Hourglass deformity,
* Circumferential plaque,
* Septal or ventral plaque,
* Plaque that cannot be palpated during clinical examination,
* Previous intralesional injection for Peyronie's Disease,
* Severe erectile dysfunction (EHS < 3),
* Current penile, malignancy,
* Previous penile surgery except for circumcision or condyloma removal,
* Previous pelvic radiation therapy,
* Anti-coagulant medication, except acetylsalicylic acid up to 100mg daily,
* Previous low-intensity focused shockwave therapy on penis,
* Any other condition that would prevent the patient from completing the study, as judged by the principal investigator,
* Being deprived of liberty or under guardianship.

Min Age: 18 Years | Sex: Male | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 120 (Actual)
Dates: Start 2021-04-06 (Actual); Primary Completion 2024-05-24 (Actual); Study Completion 2024-05-24 (Actual)

PRIMARY OUTCOMES:
Effect of low intensity ESWT on penile curvature in erection in patients with Peyronie's disease | 15 months
  Average change in penile curvature based on the pictures taken by the patient (face and profil) at baseline and after the 6 week follow-up.
  The assessment will be performed by a blinded assessor at the end of the study

SECONDARY OUTCOMES:
Assessment of the safety of ESWT on patients with PD: adverse events | 3 months
  Treatment related adverse events recorded at each visits.
Assessment of the effect of ESWT on penile pain | 3 months
  Patient complete at each visit a numeric rating scale of penile pain graduated from 0 (no pain) to 10 (worst pain) 0 means the patient has no pain and 10 for worst pain
Assessment of the effect of ESWT on sexual bother | 3 months
  Difference of the score of the International Index of Erectile Function (IIEF-5) reported by the patient at baseline and after 6 week follow-up.
  The score is calculated through 5 questions with answers ranging from 0 to 5. Between 26 and 30, the score indicates no erectile dysfunction. Between 17 and 25, it indicates mild dysfunction. Between 11 and 16, it indicates a moderate dysfunction and below 10 a complete or severe dysfunction.

CONTACTS AND LOCATIONS:
Overall Officials: Thierry LEBRET, PhD, Principal Investigator — Hopital Foch
Locations (4):
- France (4):
  - Centre d'Urologie du Polygone, Montpellier
  - Hôpital Pasteur 2, Nice
  - Foch hospital, Suresnes
  - Hôpital Rangueil, Toulouse

IPD SHARING:
Plan to Share IPD: No